CLINICAL TRIAL: NCT06163716
Title: GOIZ ZAINDU Trial: a FINGER-like Multidomain Lifestyle Intervention Feasibility Study to Prevent Dementia in Southern Europe.
Brief Title: GOIZ ZAINDU Feasibility Multi Domain Trial to Prevent Dementia.
Acronym: GOIZ_ZAINDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion CITA-alzheimer (Other)
Collaborators: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Principal Investigator, Mikel Tainta, MD, Fundacion CITA-alzheimer
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GZ trial
Record Dates: First submitted 2023-11-23; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Decline; Dementia Risk Factors; Prevention; Multidomain Intervention
Keywords: Cognitive decline; Dementia prevention; Lifestyle; Multidomain intervention; Randomized trial
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The GOIZ ZAINDU pilot trial is a one-year controlled, randomized, multidomain intervention trial, for prevention of cognitive decline, carried out in the municipality of Beasain in the Basque Country (Spain).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular health advice control (RHA) group. (No Intervention): Participants randomized to the control group followed preventive programs already ongoing at their Primary Care Unit regarding physical activity, socialization, and smoking and alcohol usage. Visits to the GP and nurse depended on personal demands and necessities; nevertheless, annual consultation was recommended for all patients over 60 years old.
- Multidomain intervention (MD-Int) group (Experimental): The MD-Int program was designed to provide tools and routines that participants could incorporate into daily living activities and reinforce the social environment. Although the program included standardized guidelines and exercises, each participant was considered individually, adapting nutritional requirements and physical and cognitive activity according to individual needs and abilities. This methodology is based on the FINGER trial design but has been adapted to local resources and the healthcare system. GPs and nurses were involved in the follow-up visits. Most intervention activities were carried out at the local Primary Care Centre. Local town hall resources such as group activities for older adults at the municipality sports centre and current outdoor sports activities were incorporated in the study.
  Interventions: Behavioral: Multidomain intervention (MD-Int) group

INTERVENTIONS:
Behavioral: Multidomain intervention (MD-Int) group — The MD-Int program included: 1) individual follow-up visits every three months for cardiovascular risk factor monitoring and nutritional counselling with primary health care providers; 2) two nutritional workshops led by a nutritionist; 3) 20 hours of cognitive stimulation delivered through group sessions and 4) 40 hours of individual cognitive training exercises. Participants in the MD-Int group received recommendations to practice 2 to 6 hours of physical exercise per week and get involved in sports activities. Social stimulation was promoted through group activities.
  Arms: Multidomain intervention (MD-Int) group

SUMMARY:
GOIZ ZAINDU ("caring early" in Basque) is a pilot study to adapt the Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER) methodology to the Basque population and evaluate feasibility and adherence to a FINGER-like multidomain intervention program. Additional aims included the assessment of efficacy on cognition and collecting data to design a large efficacy trial.

DETAILED DESCRIPTION:
The GOIZ ZAINDU pilot trial is a one-year controlled, randomized, multidomain intervention trial, for prevention of cognitive decline, carried out in the municipality of Beasain in the Basque Country (Spain). Participants were recruited in collaboration with the primary care center health providers from Beasain Municipality after an informative prevention campaign on lifestyle and dementia.

After the baseline evaluation, all participants received in person verbal information on the potential benefits of caring for vascular risk factors, adhering to Mediterranean diet, and having good cognitive and physical activity routines. Participants were later randomly assigned to a standard health advice control group (RHA, control) or the multidomain intervention group (MD-Int). Random assignment followed a proportion of 1:1 and was stratified by age (<75 years vs.≥75 years), sex, and cognitive status (normal cognition vs. MCI).

1. Regular health advice control (RHA) group. Participants randomized to the control group followed preventive programs already ongoing at their Primary Care Unit regarding physical activity, socialization, and smoking and alcohol usage. Visits to the GP and nurse depended on personal demands and necessities; nevertheless, annual consultation was recommended for all patients over 60 years old.
2. Multidomain intervention (MD-Int) group. The MD-Int program was designed to provide tools and routines that participants could incorporate into daily living activities and reinforce the social environment. Although the program included standardized guidelines and exercises, each participant was considered individually, adapting nutritional requirements and physical and cognitive activity according to individual needs and abilities. This methodology is based on the FINGER trial design[23] but has been adapted to local resources and the healthcare system. GPs and nurses were involved in the follow-up visits. Most intervention activities were carried out at the local Primary Care Centre. Local town hall resources such as group activities for older adults at the municipality sports centre and current outdoor sports activities were incorporated in the study. The MD-Int program included: 1) individual follow-up visits every three months for cardiovascular risk factor monitoring and nutritional counselling with primary health care providers; 2) two nutritional workshops led by a nutritionist; 3) 20 hours of cognitive stimulation delivered through group sessions and 4) 40 hours of individual cognitive training exercises. Participants in the MD-Int group received recommendations to practice 2 to 6 hours of physical exercise per week and get involved in sports activities. Social stimulation was promoted through group activities.

ELIGIBILITY:
Inclusion Criteria:

* Participants were at least 60 years of age,
* had a CAIDE score ≥ 6 points and
* performed below than expected in at least one of two brief cognitive tests - Memory alteration test (T@M) and Fototest
* or scored two or higher in the AD8 informant's questionnaire of cognitive symptoms.

Exclusion Criteria:

* Exclusion criteria included the presence of poorly controlled cardiovascular or respiratory disease,
* previous diagnosis of dementia, ongoing neurological disorders, unstable psychiatric disease, evidence of any other severe disease of any etiology,
* or any situation, in the investigator's opinion, that could compromise safe engagement in the intervention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Retention rate | up to 1 year
  Retention rate was defined as the proportion of participants who completed the 12-month trial period. We considered a successful rate if less than 20% of participants dropped out.
Adherence to each intervention component | up to 1 year
  Study coordinators assessed the adherence to intervention activities by recording the number of workshops and follow-up visits attended and by checking the cognitive training workbook. Self-reported information on weekly physical activity and attendance to group activities at the sports center was recorded for physical exercise.

SECONDARY OUTCOMES:
Global Cognitive performance | up to 1 year
  Cognitive performance was assessed at baseline and 12 months with the modified Neuropsychological Test Battery (NTBm) which includes the following test: Wechler Memory Scale-III Logical Memory, Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List, WMS-R Visual Paired Associates, Category Fluency, Wechler Adult Inteligence Scale-III Digit Span, Concept Shifting Test, Trail Making Test, a shortened 40-stimuli version of Stroop Test, and Letter Digit Substitution Test.
Performance in each cognitive domain | up to 1 year
  NTBm Cognitive global, executive function, memory, processing speed scores will be obtained. Composite cognitive z-scores based on the results from all single tests will be calculated. Single z-scores will be calculated using baseline mean and standard deviations of the study sample and, for each composite score, single z-scores will be averaged. Higher scores suggest better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Tainta, MD, Principal Investigator — Study Principal Investigator; Pablo Martinez-Lage, MD, PhD, Study Chair — Scientific Director
Locations (1):
- CITA-alzheimer, Donostia / San Sebastian, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: Yes
Consent for publication. All participants signed the corresponding informed consent which included an explicit consent for publication the study results and experience.
  Availability of data and materials. The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Derived] Tainta M, Ecay-Torres M, de Arriba M, Barandiaran M, Otaegui-Arrazola A, Iriondo A, Garcia-Sebastian M, Estanga A, Saldias J, Clerigue M, Gabilondo A, Ros N, Mugica J, Barandiaran A, Mangialasche F, Kivipelto M, Arrospide A, Mar J, Martinez-Lage P; GOIZ ZAINDU study group. GOIZ ZAINDU study: a FINGER-like multidomain lifestyle intervention feasibility randomized trial to prevent dementia in Southern Europe. Alzheimers Res Ther. 2024 Feb 27;16(1):44. doi: 10.1186/s13195-024-01393-z. PMID 38413990